CLINICAL TRIAL: NCT06018649
Title: The Effectiveness and Safety of Using Lithuania's Natural Resources to Improve Stress-related Mental and Physical Health
Brief Title: The Effectiveness of Natural Resources for Reducing Stress
Acronym: LUGISES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Klaipėda University (Other)
Collaborators: Research Council of Lithuania (Other)
Responsible Party: Principal Investigator, Lolita Rapoliene, Associate professor dr., Klaipėda University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BE-2-87
Record Dates: First submitted 2023-08-19; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Distress, Emotional; COVID-19
Keywords: stress; balneotherapy; mineral water; peloids; mental state; cortisol; rehabilitation; spa therapy; hydrotherapy; nature therapy; resort medicine; health; natural resources
MeSH Terms: conditions — COVID-19 | interventions — Balneology

STUDY DESIGN:
Intervention Model Description: In a parallel study 6 groups of participants will receive different interventions modalities (duration, procedures complex, inpatient/outpatient, control). Participants will be assigned to one of the treatment arms at the beginning of the trial and continue in that arm throughout the length of the trial. Assignment to a group will be randomized. There will be possibility to compare few treatments modalities results.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The subject will be randomly assigned to the study group (I-VI) by a computer program after the initial examination (T0) at the study centers. Grouping will be done by a statistician. Coding/blinding will be done so that researchers, statisticians, etc. will not know which group the subject belongs to. After the initial screening, the completed questionnaires will be modally coded by a statistician. The researchers conducting the clinical trial will not know which group the subject belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Short ambulatory balneotherapy (SAB) (Experimental): Group I will be given a complex of balneological procedures: swimming pool 20 min, 34-36° mineral/geothermal water procedure 20 min, sapropel wrapping 20 min, salt therapy 25 min. Duration of treatment - 6 days, outpatient.
  Interventions: Combination Product: Balneotherapy plus complex
- Long ambulatory balneotherapy (LAB) (Experimental): Group II will be given a complex of balneological procedures as group I- swimming pool 20 min, 34-36° mineral/geothermal water procedure 20 min, sapropel wrapping 20 min, salt therapy 25 min.
  Duration of treatment - 11 days, outpatient treatment.
  Interventions: Combination Product: Balneotherapy plus complex
- Combined nature resources treatment (CNT) (Experimental): Group III will be given a complex of balneological procedures like groups I and II plus natural therapy procedure developed by the researchers: a 45-minute walk in nature (forest, seaside), a complex of simple strength and breathing low-intensity exercises, sensory impulses (landscape , forest smells - aromatherapy, natural sounds of nature, collecting nature's goodies (berries, pine cones, leaves, etc.), awareness therapy, heliotherapy.
  Duration - 11 days., outpatient treatment.
  Interventions: Combination Product: Combined nature resources treatment
- Long inpatient balneotherapy (LIB) (Experimental): Group IV will be accommodated in the research/resort center and will receive balneological treatment (as groups I and II).
  Duration of treatment 11 days, inpatient treatment.
  Interventions: Combination Product: Balneotherapy plus complex
- Nature therapy (NT) (Active Comparator): Group V will be given only the natural therapy procedure (as in group III). Duration 11 days, outpatient, self-managed according instructions and training provided.
  Interventions: Other: Nature therapy procedure
- Control (No Intervention): Group VI - the control group, the participants of which will not be given any procedures. Duration 11 days.

INTERVENTIONS:
Combination Product: Balneotherapy plus complex — The three groups of study (SAB, LAB, LIB) will get same balneotherapy intervention with the difference in duration and mode (outpatient/inpatient). Balneotherapy plus complex procedures: swimming pool with light exercises- 20 min (29-31°C), rest 15 min, wrapping/bath with peloids (peat mud, sapropel)- 20 min (38-40°C), rest 20 min, mineral water bath- 20 min (36-38°C), salt therapy- 25 min (humidity 35%, temperature about 22°).
  Arms: Long ambulatory balneotherapy (LAB); Long inpatient balneotherapy (LIB); Short ambulatory balneotherapy (SAB)
Combination Product: Combined nature resources treatment — The participants of CNT group will be given combined treatment: nature therapy procedure (45 min) and balneotherapy plus complex intervention procedures.
  The nature therapy procedure was created by researchers by combining the principles of nature therapy, mindfulness, wild nature therapy, kinesiology selecting actions suitable for the season. A procedure instructions with specific steps will be prepared and given to the research participant. The procedure will be performed for the first time by a physiotherapist, the rest of the procedures are performed independently, following the detailed procedure with written instructions given to the participants. Each day participants will receive a message with a reminder to perform the natural therapy procedure. Duration of procedure- 45 min, outside (seaside, forest).
  Arms: Combined nature resources treatment (CNT)
Other: Nature therapy procedure — The participants of NT group will be given nature therapy procedure (45 min) created by researchers by combining the principles of nature therapy, kinesiology, mindfulness, wild nature therapy, selecting actions suitable for the season. A procedure instruction with specific steps will be prepared and given to the research participant. The procedure will be performed for the first time by a physiotherapist, the rest of the procedures are performed independently, following the detailed procedure with written instructions given to the participants. Each day participants will receive a message with a reminder to perform the natural therapy procedure. Duration of procedure- 45 min, outside (seaside, forest).
  Arms: Nature therapy (NT)

SUMMARY:
High levels of stress cause serious health problems and reduce the quality of life. There is a lack of research proving the use of natural resources for the treatment or prevention of the stress and recovery from post Covid-19 condition. The goal of research: to assess the impact of natural resources (geothermal/mineral water, mud, salt, climate) on reducing stress and improving stress-related mental and physical health, as well as the safety of the procedures. The study will be randomized, controlled, parallel group, single- blinded (to researchers). The complex of procedures of water pool, mineral water bath, mud wrapping, salt therapy, nature therapy procedure will be provided with the different duration and mode (inpatient, outpatient). Primary outcomes- the effect on stress level; secondary outcomes: the effects on stress-related mental and physical health, work and social adaptation, tolerance and safety of balneotherapy procedures. The observation: before, after treatment, after 3 and 6 month of follow-up will be reveled.

DETAILED DESCRIPTION:
The burden of stress and the consequences of Covid-19 pandemia complicates the existing capacities of the health care system and harms the efficiency and economy, therefore effective strategies are needed to reduce the consequences by creating science-based methodologies to strengthen and restore health in resorts, which would encourage wellness services, using the unique natural resources available in Lithuanian resorts and resort areas, development and would allow to compete with the most advanced European health and rehabilitation centers.

Objectives of biomedical research:

1. To assess the effectiveness of Lithuania's unique natural resources in reducing stress and improving stress-related mental and physical conditions.
2. After identifying the group of those who have recovered from Covid-19, evaluate the effectiveness of natural factors for improving this condition.
3. To present methodological recommendations for the use of Lithuania's natural resources.

Hypotheses of biomedical research:

1. It is likely that a complex of procedures using natural resources will reduce stress, anxiety, and depression.
2. It is likely that procedures with nature factors improve work and social adaptation.
3. The effect of natural resource therapy is effective regardless of the duration of treatment and season.

A multicenter, prospective, randomized controlled, single-blinded parallel group scientific study will be made.

Participants: 330 participants experiencing increased and poorly controlled stress or reduced sense of well-being in Klaipėda and Druskininkai territories (6 groups of 55 people each). Sampling is a probabilistic nest (cluster), in which each research participant's entry into the sample is multi-stage, criterion-referenced. The sample size required for statistically significant comparisons of the rehabilitation effect of the means of quantitative variables before and after the procedures was calculated by the G*Power program.

* The subject will be randomly assigned to the respective group (I-VI) by a computer program after the initial examination (T0) at the study centers. Grouping will be done by a statistician.
* • coding/blinding (if applicable, a description is provided so that no one (subjects, researchers, statisticians, etc.) will know which group the subject belongs to),
* After the initial screening, the completed questionnaires will be modally coded by a statistician. The researchers conducting the clinical trial will not know which group the subject belongs to.

Group I will be given a complex of balneological procedures: swimming pool 20 min, 34-36° mineral/geothermal water procedure 20 min, sapropel wrapping 20 min, salt therapy 25 min. Duration of treatment - 6 days.

Group II will be given a complex of balneological procedures as group I. Duration of treatment - 11 days. Comparing the results of groups I and II will allow us to assess the influence of treatment duration.

Group III will be given a complex of balneological procedures like groups I and II and a natural therapy procedure developed by the researchers: a 45-minute walk in nature (forest, seaside), a complex of simple strength and breathing low-intensity exercises, sensory impulses (landscape , forest smells - aromatherapy, natural sounds of nature, collecting nature's goodies (berries, pine cones, leaves, etc.), awareness therapy, heliotherapy.Duration - 11 days. Comparison of groups I and II will allow to evaluate the influence of complex treatment, including nature therapy.

Group IV will be accommodated in the research center and will receive balneological treatments (as groups I and II). Duration of treatment 11 days. Comparison of the effect between groups I, II, III and IV will allow to assess the impact of inpatient rehabilitation treatment relatively.

Group V will be given only the natural therapy procedure (as in group III). Duration 11 days The results will make it possible to evaluate the benefits of the natural therapy procedure, which can be applied by the person himself to improve or restore health. Comparison with the results of group II will allow to evaluate the benefits of treatment with balneotherapy procedures in the institution.

Group VI - the control group, the participants of which will not be given any procedures. Duration 11 days Comparison with groups II, IV, V will allow us to evaluate the differences in the health effects of rehabilitation procedures and natural therapy compared to no treatment.

During the study, the sociodemographic, clinical, health, body condition and safety assessment data of the study participants will be collected. Data will be collected based only on the information provided by the participant and the results obtained during the study. The screening questionnaire will ask for gender, age, marital status, education, place of residence, nature of work, length of service and earnings, information on the occurrence of Covid-19 and the incidence of chronic diseases, lifestyle habits, the level of stress experienced and methods of management, the sense of well-being experienced and information , which is important when including in the study - the current exacerbation of a chronic disease; morbidity from an oncological or infectious disease, severe form of cardiovascular, nervous, mental, kidney disease or bleeding, recent surgery or major trauma, limitation of movement function; possible pregnancy or breastfeeding; Intolerance of balneotherapy treatment or thermal procedures applied during the 3-month period and plans to leave in the next 6 months, which would not ensure your participation in the entire study period.

During the study, objective measurements will be performed to determine the response of various body systems: BP (blood pressure), HR (heart rate), SpO2 (pulsoxymetry), spirometry, toe-to-floor distance, sit-to-reach test, dynamometry, body composition analysis, waist circumference, salivary cortisol, cognitive test set (alertness, working memory, spatial number search, logical reasoning). The results of the scales will be used to evaluate the results of the study: for stress - the perceived stress scale (PSS) and the General Distress Symptoms Scale (GSDS), for anxiety - the Anxiety and Restlessness Inventory (STAI), for depression - the Center for Epidemiological Research Revised Depression Scale (CESD-R-20), for fatigue - Multidimensional Fatigue Inventory (FAS), for sleep - one-point sleep quality scale (SQS), for adaptation - Work and Social Adaptation Scale (WSAS), for well-being - Arizona Integrative Outcomes Scale (AIOS), for general health and well-being - health questionnaire, procedures security assessment questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 65 years
* Strength of stress >3 (0 no stress - 10 unbearable stress, VAS) AND/OR
* Stress control <7 (0- I can't control - 10- I control perfectly, VAS)

Exclusion Criteria:

* Uncontrolled/decompensated systemic diseases (hematological, endocrine, rheumatological, renal, cardiovascular, digestive, pulmonary),
* Active infection,
* Malignant tumors,
* Surgery or major trauma in the past year,
* Impaired ability to walk,
* Applied balneotherapy treatment during a 3-month period,
* Pregnancy/lactation,
* Bleeding,
* Severe mental disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
General Symptom Distress Scale (GSDS) | 6 month
  The GSDS is a brief self-reported measure to assess intensity (0 (I don't have this symptom) - 10 scale (extremely bothersome) of specific symptoms relevant to stress. In the second section of the GSDS, participants are asked to provide a global rating of how distressing their symptoms are on a 10-point scale, with higher scores indicating more distress. In the third part, participants are asked to provide a global rating of how well they are able to manage their symptoms on a 10-point scale with higher scores indicating better ability to manage symptoms.
PSS-10 (Perceived Stress Scale) | 6 month
  It is a self-reported questionnaire to measure the degree to which situations in one's life. There are described 10 items which are appraised as stressful and participant should sign 1-4 points to each. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. ► Scores ranging from 0-13 would be considered low stress. ► Scores ranging from 14-26 would be considered moderate stress. ► Scores ranging from 27-40 would be considered high perceived stress.
Cortisol level in saliva | Treatment (1- 2 weeks)
  Specified amount of saliva is taken into dispenser and the amount of cortisol in it is tested in sertified laboratory (Germany). Higher cortisol numbers indicate higher stress levels.

SECONDARY OUTCOMES:
Anxiety by STAI-5- Spielberger State-Trait Anxiety Inventory | 6 month
  The five-item short forms of STAIS and STAIT are given. A number of statements which people have used to describe themselves are given for the signing answer which seems to describe respondent's present feelings best. For STAIS- HOW YOU FEEL RIGHT NOW, for STAIT- HOW YOU GENERALLY FEEL in 1-4 score, where 1 means Not at all, 4- Very much so. Cutoff scores for state STAIS (>9.5) and trait STAIT(>13.5) anxiety.
Work and social adjustment by WSAS (work and social adjustment scale) | 6 month
  The effect will be measured by WSAS (work and social adjustment) scale
The safety of balneotherapy | After treatment (1-2 weeks)
  A questionnaire with 24 symptoms (redness, itching, dryness, infection, peeling, rash, red eyes, dizziness, pain, depression, insomnia, fatigue, stress, terminal pain, nausea, loss of appetite, heart palpitations, increase in blood pressure, decrease , thirst, cough, shortness of breath, general deterioration of health, and others (for enquiry) will be given to to express undesirable effects during water, mud and salt procedures. The respondent in the table indicates 1- never, 2- rarely, 3- often, 4- always, 5- required treatment. At the end participant generally assess the safety of all balneotherapy procedures at 5-point Likert scale, where 1 is very safe, 5- unsafe.
Effect on depression- CESD-R (Center for Epidemiological Studies Depression Scale ) | 6 month
  It is a 20-item measure of depressive symptoms. The list with 20 items identifies how respondent may be feeling or behaving recently. They need to check the boxes that apply how many times he have felt this way in the past week or longer. 1- Not suitable at all or Less than 1 day, 2- 1-2 days, 3- 3-4 days, 4- 5-7 days, 5- almost every day for two weeks. Bigger number means more severe depression.
Effect on fatigue- FAS-10 (Fatigue scale) | 6 month
  The scale has 10 items. Each FAS question is answered using a five-point Likert-type scale ranging from 1 ("never") to 5 ("always"). Points 4 and 10 are evaluated in contrast. The total score can range from 10, indicating the lowest level of fatigue, to 50, indicating the highest.
AIOS (Arizona Integrative Outcomes Scale) | 6 month
  AIOS scale (Arizona Integrative Outcomes Scale is a single-item visual analog scale (AIOS) where the items self-rate the overall sense of spiritual, social, mental, emotional, and physical well-being over the past 24 hours or the past month. Respondent Mark the line below with an X at the point that summarizes your overall sense of well-being for the past 24 hours from Worst you have ever been to best you have ever been.
Sleep quality | 6 month
  SQS (Single-Item Sleep Scale (Snyder E, 2018). This is a single-item sleep quality scale. The SQS is easily self-administered administered a questionnaire that uses a visual analog scale.The questionnaire instructions instruct the respondent to rate overall sleep quality over a 7-day period on a VAS from 0 to 10 based on the following five categories: 0 = terrible, 1-3 = poor, 4-6 = fair, 7- 9 = good and 10 = excellent When assessing sleep quality, respondents are asked to consider the following key components of sleep quality: how many hours they slept, how easily they fell asleep, how often they woke up during the night (except for going to the bathroom), how often they woke up earlier than they should, and how rested felt after sleep.
Cognitive function | 6 month
  Cognitive function will be measured using licenced RehaCom software screening tests (working memory, attention, working speed, attention span). Bigger positive results means better function, negative results- bad function.
Forced vital capacity | 6 month
  FVC-Forced vital capacity- the total volume of air that can be exhaled during a maximal forced expiration effort measured in litres.
Forced expiratory volume | 6 month
  The forced expiratory volume in 1 second (FEV1) is the volume of air (in liters) exhaled in the first second during forced exhalation after maximal inspiration.
Peak expiratory flow | 6 month
  PEF is measured during routine spirometry. Peak expiratory flow (PEF) is given in litres of air breathed out per minute (l/min).
Blood pressure | 6 month
  Measuring systolic and diastolic blood pressure (mmHg)
Heart rate | 6 month
  Heart rate in times per minute
Oxygen saturation | 6 month
  Using a pulse oximeter we will measure oxygen saturation. It is a noninvasive device placed over a person's finger. It measures light wavelengths to determine the ratio of the current levels of oxygenated hemoglobin to deoxygenated hemoglobin.
Skin condition | 6 month
  Skin condition will be measured: moisture, oiliness, elasticity (TMISHION Skin Tester, Model: M-6602). Portable Instrument Skin Oil Content Moisture Analyzer will measure skin moisture, oiliness, elasticity degree using bio-resistance technology which can accurately detect the health value of the skin, further understand the skin condition. The inductive probe can sense the skin condition, and can monitor the degree of whitening, moisture, oil content and skin elasticity. Higher degree indicate higher parameter measured.

CONTACTS AND LOCATIONS:
Overall Officials: Lolita Rapoliene, ass.prof., Principal Investigator — Klaipėda University
Locations (1):
- Klaipėda university, Klaipėda, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided
Sharing of participant data is possible by separate agreement, only for scientific purposes in the relevant field.